CLINICAL TRIAL: NCT05066152
Title: The Effects of Single Probiotic on Glycemic Control, Lipid Profile, Some of Inflammatory Cytokines and Gene Expression Levels in Type 2 Diabetic Patients
Brief Title: The Effect of Single Probiotic on Metabolic Control in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Beyza Eliuz Tipici, Dietician, Ph.D., Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulU-BTipici-001
Record Dates: First submitted 2021-09-14; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Lactobacillus GG; probiotic; gene expression
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: prospective, single center, interventional
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): For 8 weeks of interventional period, the patient received 10 probiotic drops (1x1010 Cfu LGG) once daily at breakfast.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG (ATCC 53103)
- Placebo (Placebo Comparator): For 8 weeks of interventional period, the patient received 10 probiotic drops (placebo) once daily at breakfast.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG (ATCC 53103) — One probiotic drop contained a formulation of 1x109 Cfu Lactobacillus rhamnosus GG (LGG; ATCC 53103)
  Arms: Probiotic
Dietary Supplement: Placebo — Carrier material of probiotic product, not containing bacterial strain, similar appearance as the probiotic
  Arms: Placebo

SUMMARY:
Recent studies indicate that dysbiosis of intestinal microbiota and low grade inflammation are important pathogenic determinants of type 2 diabetes (T2DM), which has increased in epidemic size over the last 20 years. Probiotics have been used in T2DM for the modification of IM and anti-inflammatory effects. However, effect of probiotics on metabolic control in T2DM are inconsistent.

Present study will be designed to determine the effects of Lactobacillus GG (LGG) on glycemic control, lipid profile, inflammation parameters and expression of certain genes linked to T2DM. This study will be conducted at the Istanbul Faculty of Medicine, a tertiary care diabetes outpatient clinic and should involve 34 T2DM subjects. Subjects will be randomly assign to receive either LGG probiotic drop or a placebo.In this placebo controlled trial, effect of single strain probiotic vs. placebo on metabolic control and certain genes linked to T2DM will be assessed.

DETAILED DESCRIPTION:
Evidence-based data showed that intestinal microbiota (IM) plays a role in the development of metabolic diseases. Recent studies have reported that dysbiosis of IM and low-grade inflammation is effective in pathogenesis of type 2 diabetes mellitus (T2DM), which has increased in epidemic size over the last 20 years. Firmicutes, Bacteroidetes and Proteobacteria's ratios in obese and T2DM patients were found to be different than healthy subjects. In these cases, there is an association between increasing the proportion of gram-negative bacteria in the intestines and subclinical inflammation.

Probiotics are live microorganisms that are intended to have health benefits by regulating mucosal and systemic immunity, when consumed as a nutritional supplement. There are studies investigating the effects of probiotic use on insulin sensitivity, glycemic control, lipid profile and inflammatory parameters in patients with T2DM. However, several probiotic strains were used frequently in these studies, or probiotics and prebiotics were given as cocktails. Their effects might be together or even synergistic. Lactobacillus rhamnosus GG (or Lactobacillus GG: LGG) is a widely used probiotic microorganism. Studies have shown that LGG prevents diarrhea and atopic dermatitis, provides antitumor activity, improves the immune system, and lowers serum cholesterol levels. However, there is a limited data about the effects of LGG on the glycemic control of diabetic animal models but human studies are scarce.

Therefore, present study is designed to determine the effects of LGG on glycemic control, lipid profile, inflammation parameters, and expression of certain genes linked to T2DM.

Subjects will be randomly assign to receive probiotic "Lactobacillus Rhamnosus GG (ATCC 53103)" or placebo for 8-weeks administered as a drop formulation. Patients in the intervention group receive 10 probiotic drops (1x1010 cfu LGG) once daily with breakfast. Subjects will be contacted via telephone every week for an assessment of adverse events and probiotic/placebo compliance. Fasting blood samples will be taken at baseline and post treatment to measure carbohydrate metabolism (glucose, insulin, fructosamine and HbA1c), lipid profile (triglycerides; total, HDL- and LDL-cholesterol) and biomarkers of inflammation (hs-CRP and IL-6). TLR2, TLR4, MUC2 and MUC3A genes expressions will be investigated on stool samples at baseline and post treatment. Stool samples will be stored at -80°C until RNA isolation.The gene expression levels will be determined by Quantitative Real Time PCR method using the determined cDNA samples. Dietary intake will be evaluated by the 3-day food record. During the 4th and 8th week of the study, a 3 day food consumption records will be taken. Diabetics will be given detailed oral and written instructions regarding the completion of food record, consisting of 2 midweek days and 1 weekend day. In order to determine the amounts of consumed foods correctly, information will be given about measuring cups such as water glass, tea glass, teaspoon, tablespoon, serving spoon, bowl. Dietary intake will be assessed using a food composition database of BEBIS programme including specific Turkish foods. All anthropometric measures will be conducted in a fasting state taken at baseline and following an 8-week intervention by experienced examiner (dietitian). Body weight and body composition will be assessed by bioelectrical impedance analysis device (Tanita BC-420 MA). Body mass index (BMI) will be calculated as weight (kg) divided by height squared (m2). Waist circumference (measured midway between lowest rib and iliac crest) will be measured using a non-stretchable measuring tape.

All analysis will be performed using the Statistical Package for Social Sciences (SPSS) 21.0 package program and significance will defined as p<0.05. Descriptive statistics will be given as mean, standard deviation and median (minimum to maximum) for continuous measures. Categorical variables will be expressed as case numbers and percentage values. The Shapiro-Wilk tests will used to determine whether the distribution of continuous measures are normal. Student's t test and Mann-Whitney-U test will used for the two groups comparisons according to whether the variables showed normal distribution. Comparisons of changes in groups within themselves (before and after probiotic or placebo administration) will made using the t-test if the variances is normal, and if the Wilcoxon test is not normal in the cohort. The web-based RT2 Profiler PCR Array Data Analysis program will used to determine the change of ΔCt values obtained from the Real Time-PCR gene expression study (before and after probiotic and placebo administration). p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes
* Taking oral-antidiabetic medication

Exclusion Criteria:

* Smokers,
* Alcohol drinkers,
* Inflammatory bowel or autoimmune disease,
* Immunodeficiency,
* Using anti-epileptic, incretin enhancer (DPP-4 inhibitor), insulin or insulin analogs, dietary supplements
* Systemic antibiotics within 6 weeks before inclusion
* Use of probiotics within 3 months before inclusion
* Breast-feeding or pregnancy

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | 8 weeks compared to baseline
  HbA1c %
HOMA-IR | 8 weeks compared to baseline
  HOMA-IR= Fasting plasma glucose (mg/dL) x Fasting plasma insulin (μU/mL)/405

SECONDARY OUTCOMES:
QUICKI | 8 weeks compared to baseline
  1/ [log (fasting plasma insulin (μU/mL)+log (fasting blood glucose (mg/dL)] [22, 23].
Fasting plasma glucose | 8 weeks compared to baseline
  FPG in mg/dL
Fructosamine | 8 weeks compared to baseline
  μmol/L
HDL-C | 8 weeks compared to baseline
  mg/dl, HDL cholesterol
LDL-C | 8 weeks compared to baseline
  mg/dl, LDL cholesterol
Triglycerides | 8 weeks compared to baseline
  mg/dl
hs-CRP | 8 weeks compared to baseline
  mg/dl, high sensitive c reactive protein
IL-6 | 8 weeks compared to baseline
  pg/mL, Interleukin 6
TLR2 | 8 weeks compared to baseline
  Toll-like receptor 2 gene expression
TLR4 | 8 weeks compared to baseline
  Toll-like receptor 4 gene expression
MUC2 | 8 weeks compared to baseline
  Mucin 2 gene expression
MUC3A | 8 weeks compared to baseline
  Mucin 3A gene expression
Weight | 8 weeks compared to baseline
  body weight, kg
BMI | 8 weeks compared to baseline
  body mass index, kg/m2
WHR | 8 weeks compared to baseline
  waist and hip ratio %
Fat mass | 8 weeks compared to baseline
  body fat mass, kg
Fat mass | 8 weeks compared to baseline
  body fat mass, %
Lean body mass | 8 weeks compared to baseline
  body lean body mass, kg
Muscle mass | 8 weeks compared to baseline
  body muscle mass, kg
Total body water | 8 weeks compared to baseline
  kg kg and %
Total body water | 8 weeks compared to baseline
  % kg and %
Bone mass | 8 weeks compared to baseline
  Body bone mass, kg
Basal metabolic rate | 8 weeks compared to baseline
  Acoording to bioelectrical impedance analysis device, kcal
Energy | During 4th and 8th weeks
  Energy intake, kcal
Carbohydrate | During 4th and 8th weeks
  Carbohydrate intake, gram
Carbohydrate | During 4th and 8th weeks
  Carbohydrate intake, %
Protein | During 4th and 8th weeks
  Protein intake, gram
Protein | During 4th and 8th weeks
  Protein intake, %
Fat | During 4th and 8th weeks
  Fat intake, gram
Fat | During 4th and 8th weeks
  Fat intake, %
Dietary fiber | During 4th and 8th weeks
  Dietary fiber intake, gram
Dietary cholesterol | During 4th and 8th weeks
  Dietary cholesterol intake, gram

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eliuz Tipici B, Coskunpinar E, Altunkanat D, Cagatay P, Omer B, Palanduz S, Satman I, Aral F. Lactobacillus GG is associated with mucin genes expressions in type 2 diabetes mellitus: a randomized, placebo-controlled trial. Eur J Nutr. 2023 Aug;62(5):2155-2164. doi: 10.1007/s00394-023-03139-3. Epub 2023 Mar 30. PMID 36997822